CLINICAL TRIAL: NCT06092619
Title: Effects of Vojta Therapy on the Motor Function of Children With Neuromotor Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Principal Investigator: Juan Luis Sánchez González, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VojtaTherapy
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Motor Disorders
Keywords: Vojta Therapy; Neuromotor disorders; Motor function; Children
MeSH Terms: conditions — Motor Disorders

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial has been designed that will assess gross motor function from the start of the rehabilitation intervention (with Vojta therapy or other methodologies).
Who Masked: Outcomes Assessor
Masking Description: Neither the therapists nor the evaluators of the GMFM may be blinded to the type of treatment administered due to the organization of the Rehabilitation service where the study is carried out, as well as the "face-to-face" requirements for carrying out the Vojta therapy and the evaluation. of that scale. However, the assessment of the Infant Motor Profile (IMP) is performed by observing a protocolized video recording. This would allow the quantification of this escape by an evaluator external to the service (in this case the external Principal Investigator). This would allow not only to blind the evaluator regarding the type of intervention that the child receives, but also if the video belongs to pre or post intervention. To do this, the videos will be sent encrypted and randomized for quantification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients under Vojta Therapy intervention
  Interventions: Other: Vojta Therapy
- Control Group (Active Comparator): Patients under regular physiotherapy intervention
  Interventions: Other: Conventional physiotherapy:

INTERVENTIONS:
Other: Vojta Therapy — The therapist applied pressure to defined zones on the body whilst positioned in prone, supine and side lying, where the stimulus leads to automatically and involuntarily complex movement.The parents were also instructed on at least one of the exercises from the first session, after the initial assessment. The home program was progressively increased and supervised until the three therapy positions were mastered, during weekly or fortnightly follow ups. The recommended dose was four times per day at home, in session no longer than 15-20 minutes; however, the daily frequency of each family due to different availability was also taken in account. The frequency of the dose was divided into 3 groups: families who could carry on therapy a) three times per day, b) four times per day, c) one or two times per day, d) less than seven times per week or therapy at the clinic
  Arms: Intervention Group
Other: Conventional physiotherapy: — Conventional physiotherapy intervention included goal-directed functional training based on tasks. These motor skills will be performed in enhanced and adapted settings, but as similar as possible to the usual activities of daily living. Family and children participated in the goal setting, and the approach will focus on overcoming the limitations of the activities to reach these, instead of the modification of the movement patterns. This intervention is founded in motor learning and behavioral neuroscience, focusing on participation and activity acquisition.
  Arms: Control Group

SUMMARY:
Functionality and motor skills during activities of daily living have progressively gained importance as tools for classification, assessment and research of neuromotor disorders and the treatment methodology according to Dr. Vojta or Reflex Locomotion follows this criterion in the clinical field. Vojta therapy is a commonly extended tool in the field of pediatric rehabilitation. This methodology acts on the ontogenic postural function and automatic postural control, on which different environmental aspects will later act. It is not a functional training, to avoid the voluntary movement available according to the pathology by means of compensations. Vojta therapy would be the key to unlock the development of gross motor function, later used in the movement of daily life activities, including other therapies such as conventional physiotherapy, sensory stimulation, occupational therapy, etc. This study aims to demonstrate that there are changes in the motor development of children with cerebral palsy with the application of Vojta Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children
* Diagnosis of cerebral palsy or neuromotor disease

Exclusion Criteria:

* healthy subjects
* Patients receiving other therapy during the procedure

Ages: 0 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM). | Baseline and immediately after the intervention
  Gross motor function and mobility have important roles for classification, assessment and research involving children with neuromotor disorders. Gross Motor Function Measure could be currently considered as gold standard for the quantification of gross motor function in the pediatric rehabilitation. Maximum and minimum scores on the GMFM may vary depending on age and the specific dimension being assessed (0-88). In general, a score of 100% on a dimension would indicate that the child has a motor skill level equivalent to that of a nondisabled child of the same age on that dimension.
Infant Motor Profile (IMP) scale | Baseline and immediately after the intervention
  The Infant Motor Profile scale is another evidence-based method of assessing infant motor behavior. It not only quantifies motor milestones, but also movement quality by analysing five factors: variability, adaptation, symmetry, fluency, and capacity. The advantage of this scale is that the assessment is performed through video recording, allowing to have a dedicated clinical evaluator blinded to the type of intervention. There is no specific maximum or minimum IMP score value, as the scores are interpreted in relation to typical motor development skills for the child's age. In general, a higher PMI score indicates better motor development, while a lower score may suggest delays in motor development.

SECONDARY OUTCOMES:
Date of birth | Baseline
  It will be registered at the beginning of the study in order to calculate the age of the participant.
Diagnosis | Baseline
  It will be registered at the beginning of the study in order to calculate the diagnosis of the participant.
Number of previous physiotherapeutic treatments | Baseline
  Data will be collected on participants' previous treatments: Occupational Therapy; Hydrotherapy; Surgery and Botulinum toxin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menendez-Pardinas M, Alonso-Bidegain M, Santonja-Medina F, Sanchez-Gonzalez JL, Sanz-Mengibar JM. Effects of Vojta Therapy on the Motor Function of Children with Neuromotor Disorders: Study Protocol for a Randomized Controlled Trial. J Clin Med. 2023 Nov 28;12(23):7373. doi: 10.3390/jcm12237373. PMID 38068424